CLINICAL TRIAL: NCT01499875
Title: A Pharmacokinetic and Pharmacodynamic Study of Phenoxymethylpenicillin for Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Department of Microbiological Surveillance and Research, SSI. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Penicillin
Record Dates: First submitted 2011-08-18; First posted 2011-12-26 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2013-01

CONDITIONS: Phenoxymethylpenicillin
Keywords: Pharmacokinetic; Pharmacodynamic; Phenoxymethylpenicillin; Children
MeSH Terms: interventions — Penicillin V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phenoxymethylpenicillin (Other): It is a descriptive trial to find out about the pharmacokinetics
  Interventions: Drug: Phenoxymethylpenicillin

INTERVENTIONS:
Drug: Phenoxymethylpenicillin — mixture, 25 or 50 mg/kg taken once.
  Other Names: Primcillin

SUMMARY:
The aim of this trial is to evaluate the pharmacokinetics and pharmacodynamics of penicillin V in non-infectious children to estimate the optimum dosage regime in children.

DETAILED DESCRIPTION:
Although occasionally questioned, the efficacy of penicillin in eradication of respiratory tract infections in children has not been convincingly reported in the literature. Two randomized multicenter antibiotic efficacy trials have been reported in eradication of group A streptococci where both oral and intramuscular administration of penicillin had relatively high microbiologic failure rates. But the trials only confirm that the treatment is not effective in the given dose. The recent recommendations on penicillin are unfortunately based upon past practices, clinical trial results and recent resistance trends and pharmacodynamics have not been considered to support the choice of drug and dosage regimen. Some pharmacodynamic trials have been made on meropenem, cefotaxime, piperacillin-tazobactam and amoxicillin in children but so fare no trials have been described on penicillin. It is well described in adults but the absorption and secretion might be depended on age. Penicillin exhibit a time-dependent killing which means that the time over minimal inhibitory concentration (MIC) is the parameter best related to efficacy.

Methods:

The investigators evaluate the pharmacokinetics and pharmacodynamics of penicillin V in non-infectious Danish children at age 0-10 years who were admitted for a chromium-51-EDTA-clearance test. The investigators excluded children with allergy to penicillin and children with a prior known reduced glomerular filtration rate. The parents of each child who participated gave written informed consent before the study and ethical approval was obtained.

Antimicrobial dosage and administration:

40 children were assigned to receive per oral penicillin suspension 22-32 mg/kg. The dosage was estimated 25 mg/kg by the weight the parents rapported and they had a weight control at admission. The exact given dose was then calculated. The penicillin were not taken on an empty stomach to imitate reality as much as possible and the time of administration was noted. Another 40 children were given 50 mg/kg penicillin mixture.

Samples:

Blod samples of 1 ml were taken after 0, 15, 30, 60, 90, 120 minutes after the Crom-EDTA examination had started giving a dispersion in time compared to the intake of penicillin. The samples were collected in vacuum tubes containing EDTA as an anticoagulant and then centrifuged quickly. The separated serum were placed in cryovials before frozen.

ELIGIBILITY:
Inclusion Criteria:

* Non-infectious Danish children at age 0-10 years who were admitted for a chromium51EDTA clearance test

Exclusion Criteria:

* Children with allergy to penicillin and children with a prior known reduced glomerular filtration rate

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Phenoxymethylpenicillin concentrations | up to 7 hours after the penicillin is taken
  The data will be presented before June 2013

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Birkebæk, PhD, Study Chair — Department of Pediatrics, Århus University Hospital, Skejby
Locations (1):
- Department of Pediatrics, Århus University Hospital, Skejby, Aarhus, Denmark